CLINICAL TRIAL: NCT05575960
Title: Interpersonal Psychotherapy for Adolescents and Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linnaeus University (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Fredrik Falkenstrom, Professor of Clinical Psychology, Linnaeus University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022-00983
Record Dates: First submitted 2022-10-04; First posted 2022-10-12 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Intervention Model Description: Multiple Baseline Design
Masking Description: Not possible to mask psychotherapy for patient or therapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interpersonal Psychotherapy (Experimental): Interpersonal Psychotherapy for Adolescents according to the manual by Mufson (2004).
  Mufson, L. (2004). Interpersonal psychotherapy for depressed adolescents. Guilford Press.
  Interventions: Behavioral: Interpersonal Psychotherapy for Adolescents (IPT-A)

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for Adolescents (IPT-A) — Interpersonal Psychotherapy (IPT) is a psychotherapeutic treatment originally developed for treating depression in adults. It is a brief, structured treatment based on the idea of mobilizing the patient's social network, increasing his/her capacity to accept and seek support from others, and to process interpersonal difficulties, in order to improve depressive symptoms. Interpersonal psychotherapy for adolescents (IPT-A) is a version of IPT designed for young people between the age of 12-18 years with depression (Mufson, 2004), and is in many respects similar to IPT although with some modifications (e.g., a few scheduled meetings with parents during the course of treatment).

SUMMARY:
The purpose of the project is to study the effectiveness of Interpersonal Psychotherapy (IPT) for adolescents with depression. Specific aims are to analyze the effects, change mechanisms, predictors, and implementation of IPT for youth. In this four-year project we will include 60 patients with depression. Outcome will be studied using a quasi-experimental multiple-baseline design. Change mechanisms will be studied in the form of mentalizing, emotion regulation, social support, and working alliance session-by-session, and with post-treatment qualitative interviews about the participants' experiences of change. Predictors of effectiveness of IPT for adolescents will be explored by measuring severity of symptoms, anxiety symptoms, presence and severity of parent-child conflicts, quality of interpersonal relationships, experiences of bullying, and school functioning. The implementation process of IPT for youth will be studied through interviews with adolescents, parents, therapists, co-workers, and local managers.

The study is conducted within child and adolescent psychiatric services in Norrköping using a practice-oriented research strategy which emphasizes close collaboration with clinicians. The project is a collaboration between researchers at Linnaeus University and Linköping University, and clinicians at BUP Norrköping.

DETAILED DESCRIPTION:
Aim: To analyze the effects and the usefulness of IPT for adolescents with depression .

Site Norrköping Child and Adolescent Psychiatric Services BUP Norrköping receives approximately 820 new patient every year, and about 285 of these are diagnosed with depression. Seven therapists are working with IPT for adolescents. (Depression data)

Patients Inclusion and exclusion criteria will be evaluated using the Mini-International Neuropsychiatric Interview.

Therapists The requirement of therapists is to have IPT training of at least level B. All therapists will be employed within the Child and Adolescent Psychiatric Services, and work under the regulations of the Health Care Act.

Sample Size It is estimated that recruiting and treating 15-20 patients a year will be feasible. In four years, 60 adolescents with depression will be recruited.

Statistical Power Power was calculated by running Monte Carlo simulation analyses. The difference between treatment and baseline was assumed to be similar to the difference between treatment and waiting lists in between-group randomized trials, which is usually above d = 0.80. Power was evaluated for the same statistical method that will be used in outcome analysis. Assuming an effect size of d = 0.80 and a sample size of 60, statistical power for the difference between the treatment and baseline slopes was 84%.

Measurement Instruments For outcome measures, longer scales are used before starting and at the end of treatment, and shorter measures are filled out prior to each session. The process measures are used each session, and match roughly the theoretically identified IPT change mechanisms (Lipsitz & Markowitz, 2013).

Outcome Measures: Depression (i) Montgomery Åsberg Depression Rating Scale is a widely used measurement instrument for depressive symptoms. It has been validated for use with adolescents. The observer version of MADRS will be administered before waiting list, at treatment start, and at termination, using the structured interview SIGMA.

(ii) Patient Health Questionnaire - 9M is based on the DSM criteria for major depressive disorder, with nine items focusing on depressive symptoms and ask the individual to rate the duration for which they experienced each symptom. The 9M version is adjusted specifically to the diagnostic criteria for adolescent depression. Items are scored on a Likert scale of 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 27. The PHQ-9 has demonstrated high sensitivity (89.5%) and good specificity (78.8%) in detecting depression in adolescents in a care sample. The PHQ-9 will be administered before the start of each session.

Change Process Measures Rated by External Observers (i) Symptom-Specific Reflective Functioning is a measure of the capacity for understanding connections between psychiatric symptoms, mental states, and interpersonal relationships; in other words, mentalizing about psychiatric symptoms. This capacity has been postulated to be especially relevant for IPT, due to its focus on connecting symptoms with interpersonal relationships and emotions. External raters will rate SSRF from the first few minutes of each session, in which IPT therapists ask about symptoms and interpersonal relationships from the previous week.

Change Process Measures Rated by Therapists (i) Working Alliance Inventory - Short form Revised, therapist version is a 12-item measure of the quality of the working alliance, i.e., collaborative relationship, between therapist and patient. This measure is administered to therapists immediately after each session.

Change Process Measures Rated by Patients (i) Session Alliance Inventory is a six-item patient-report measure of the quality of the working alliance, i.e., collaborative relationship, between therapist and patient during the previous session. This measure is administered to both patients and therapists immediately after each session.

(ii) Brief Mentalized Affectivity Scale is a validated patient-report measure for assessing emotion regulation. The short version (12 items) will be filled out immediately before each session.

(iii) Social Support Questionnaire - 6 asks about the person's available network for social support, the availability and quality of support from the network. This will be filled out at treatment start, at mid-treatment, and at treatment termination.

Study 1: Test the Effectiveness of IPT using a Quasi-Experimental Multiple-Baseline Design.

A non-concurrent multiple baseline design will be used, that is, not all patients start treatment at the same time. The sequence will be an A1BA2 design, in which A means no treatment and B means treatment. A1 is the baseline and A2 is the follow-up period. The distinction between A1 and A2 is due to the fact that reversibility of effects in the follow-up phase are not expected. The fact that waiting times vary quasi-randomly according to availability in the therapists' calendars will be utilized, with a minimum waiting of three weeks to establish a slope for the baseline period. Data for Study 1 will be analyzed using a piecewise multilevel growth curve model, in which two separate slopes for change over time in the outcome measure - one for the baseline phase and one for the treatment phase - are compared. If treatment is effective, symptoms should improve at a faster rate during treatment than before treatment. Thus, the test is the average change rate during the treatment phase minus the average change rate during the baseline phase.

Study 2: Mechanisms of change in IPT-A for depression Longitudinal (session-by-session) observation study using data from the treatment phase (B). Specifically, the proposed change mechanisms (mentalization, emotion regulation, social support, and working alliance) are measured each session, and used to predict next-session outcome. In addition, post-treatment qualitative interviews with patients will be used to retrospectively study the participants' experiences of change and what contributed to this. For Study 3, disaggregated time-lagged panel models will be used, in which candidate mechanisms of change are used as predictors of change in the outcome measure from one session to the following session.

Study 3: Predictors of improvement in IPT-A for depression Longitudinal observation design using baseline data on patients to predict differential trajectories during the treatment- and follow-up phases to explore for which patients IPT-A is effective. Session-wise measurements will be used to enable tests of causal direction for the candidate mechanisms. Multilevel growth curve modeling using pre-treatment variables as predictors of the intercepts and slopes of the outcome measure will be used. The cross-level interaction between a pre-treatment variable and the slope of time is the test of interest. Based on previous research, severity of symptoms (depression/eating disorder), comorbid anxiety disorder, the presence and severity of parent-child conflicts, quality of interpersonal relationships, experiences of bullying, and school functioning will be explored as potential predictors of IPT effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder according to the DSM-V
* Age 15 to 17,5 years.
* Good-enough knowledge in Swedish to be able to read instructions in questionnaires and who do not require an interpreter.

Exclusion Criteria:

* Ongoing psychosis
* Drug or alcohol addiction
* Bipolar disorder
* Suspected mental retardation
* Acute suicidality or severe depression requiring hospitalization
* Patients who have started antidepressant medication within the last six weeks will need to wait until medication effects have stabilized.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire - 9 for depression/Eating Disorder Inventory - Very Short for eating disorder patients | Change from treatment start to week 12 compared to change from before waiting-list to treatment start. In the multiple baseline design, the time for the waiting list varies, in this case about 4-25 weeks.
  Patient-rated depression/eating disorder severity. Scale from 0-27 points, with higher scores indicating more severe symptoms.
Montgomery Åsberg Depression Rating Scale (observer version) for depression/Eating Disorder Inventory for eating disorders | Change from treatment start to week 12 compared to change from before waiting-list to treatment start. In the multiple baseline design, the time for the waiting list varies, in this case about 4-25 weeks.
  Depression/eating disorder severity measures. Scale from 0-60 points, with higher scores indicating more severe symptoms..

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Falkenström, PhD, Principal Investigator — Linnaeus University
Locations (1):
- Norrköping Child and Adolescent Psychiatric Services (BUP Norrköping), Norrköping, Sweden

IPD SHARING:
Plan to Share IPD: No